CLINICAL TRIAL: NCT01448070
Title: A Single Centre, Randomized, Balanced Double Blind, Cross-over Trial Investigating the Bioequivalence of Actrapid® Produced by the Current Process and Human Insulin With the Same Formulation as Actrapid®, Produced by the NN729 Process
Brief Title: Comparison of Human Insulin Produced by the Current Process and the NN729 Process in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN729-1511
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NN729 manufacturing process (Experimental)
  Interventions: Drug: human insulin
- Current manufacturing process (Active Comparator)
  Interventions: Drug: human insulin

INTERVENTIONS:
Drug: human insulin — Single dose of 0.2 IU/kg, administered subcutaneously (under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to show that the product of the new production process has a similar pharmacological profile to the traditional process used for the current commercial product Actrapid®.

ELIGIBILITY:
Inclusion Criteria:

* Normal findings in medical history and physical examination unless the investigator considers any abnormality to be clinically irrelevant
* Fasting blood glucose below or equal to 6 mmol/L
* Body Mass Index (BMI) 22.0-27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Participated in another clinical study with an investigational drug within the last 4 weeks
* Any condition requiring the regular use of any medication, including herbal remedies, over the counter medicines and vitamins. Occasional paracetamol is acceptable
* Known or suspected allergy to the trial product or related products
* Family history of type 1 diabetes

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2002-10-15 (Actual); Primary Completion 2002-12-20 (Actual); Study Completion 2002-12-20 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) 0-8h (human insulin)
Cmax (maximum plasma concentration)
Area under the curve (glucose infusion rate (GIR)), 0-8h

SECONDARY OUTCOMES:
tmax (time to reach maximum)
t½ (terminal half-life)
GIR (glucose infusion rate) max
tGIR (glucose infusion rate) max
Area under the curve (C-peptide, 0-8h)
Physical examinations and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manchester, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com